CLINICAL TRIAL: NCT01976455
Title: The Breathe Light Study: Validation of Carbon Stable Isotope Ratio in Breath as an Indicator of Energy Balance and Substrate Utilization
Brief Title: The Breathe Light Study
Status: Completed | Type: Observational
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: GFHNRC505
Record Dates: First submitted 2013-09-12; First posted 2013-11-05 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Over-eating; Obesity
Keywords: obesity; carbon13; over-eating; metabolic chamber; room calorimeter
MeSH Terms: conditions — Hyperphagia; Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 20% calorie depletion: During each 11-day stays the volunteer will have 9 days of calorie depletion (20% one stay and 40% the other).
  Interventions: Other: 20% fewer calories; Other: 40% fewer calories
- 40% calorie depletion: During each 11-day stays the volunteer will have 9 days of calorie depletion (20% one stay and 40% the other).
  Interventions: Other: 20% fewer calories; Other: 40% fewer calories

INTERVENTIONS:
Other: 20% fewer calories
Other: 40% fewer calories

SUMMARY:
The purpose of this study is to develop a novel, non-invasive method that will provide personalized feedback during dietary interventions as a marker for compliance.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* Overweight (BMI 25-40 kg/m2)

Exclusion Criteria:

* Metabolic or cardiovascular abnormalities (diabetes, uncontrolled hypertension, etc.)
* Gastrointestinal disorders
* Disease that affects macronutrient utilization
* Medication that affects macronutrient utilization
* Allergies to foods to be utilized in the study (including but not limited to lactose intolerance/milk allergy)
* Use of nutritional/sport supplements
* Pregnant or currently trying to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men & Women age 18 to 65 years with a BMI of 25- 40 kg/m2.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Increase in breath Carbon 13 with overconsumption of calories | 11 days
  A period of positive energy balance following one of negative energy balance increase breath Carbon13.

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center; James N Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No